CLINICAL TRIAL: NCT01726166
Title: A Randomized Controlled Trial: Suprapubic Aspiration Versus Urinary Catheterization in the Neonatal Intensive Care Unit.
Brief Title: Suprapubic Aspiration Versus Urinary Catheterization In Neonates.
Acronym: SPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment over 3 yrs (n=47). No chance to reach sample size (n=~160).
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Gregory Moore, Assistant Professor, Neonatologist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011813-01H
Record Dates: First submitted 2012-11-07; First posted 2012-11-14 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Neonatal Urinary Tract Infection
Keywords: Infant; contamination rates; urinary catheterization; suprapubic aspiration
MeSH Terms: interventions — Urinary Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suprapubic Aspiration (Active Comparator): A trained physician or neonatal nurse practitioner utilizing U/S guidance at the bedside will perform the SPA. An U/S machine is readily available for use in each NICU.
  Interventions: Procedure: Suprapubic Aspiration
- Urinary Catheterization (Active Comparator): The infants will have the procedure done by NICU nurses who have been trained in performing this procedure.
  If the randomly assigned infant passes urine spontaneously during a UC attempt after complete perineal cleansing and the urine is collected as a "clean catch" sample, then this infant will be analysed in the assigned group (intention to treat).
  Interventions: Procedure: Urinary Catheterization

INTERVENTIONS:
Procedure: Suprapubic Aspiration — Pain management will be performed as per our NICU protocols by administering 24% sucrose prior to both procedures to ensure adequate pain control. Additional or different analgesia may be used depending on the patient's specific clinical situation. We will use a chlorhexidine 0.05% with no cetrimide solution as the cleaning solution.
  Arms: Suprapubic Aspiration
Procedure: Urinary Catheterization — Pain management will be performed as per our NICU protocols by administering 24% sucrose prior to both procedures to ensure adequate pain control. Additional or different analgesia may be used depending on the patient's specific clinical situation. We will use a chlorhexidine 0.05% with no cetrimide solution as the cleaning solution.
  Arms: Urinary Catheterization

SUMMARY:
Urinary tract infection (UTI) is relatively common in infants, with an occurence rate of up to 10%.

Analysis of collected urine for the presence of bacteria or fungus is the only way to make a certain UTI diagnosis. Sterile collection of urine can be achieved in newborn infants by urinary catheterization (UC) where a catheter is passed through the urethra into the bladder, suprapubic aspiration (SPA) where a needle is inserted into the bladder through the abdominal wall, or 'clean catch' where urine is collected into a sterile bottle as the baby urinates during preparation for UC. The main advantage of SPA is that it bypasses the bacteria that normally resides in the urethral opening, thus minimizing the risk of contamination. Some studies have suggested that SPA is better than UC for collecting urine in a sterile fashion in the neonate due to the difficulty of doing sterile UC in small infants resulting in more contaminated samples (also called a false-positive urine culture); there is still no clear best choice. UC is commonly used in many Neonatal Intensive Care Units (NICU) as it is considered less invasive, can be done by the nursing staff, and generally has a higher chance of obtaining urine. SPA is a simple and safe alternative and, although it may be more painful than UC, it is performed more quickly. The reported success rate for SPA is variable, but is greatly increased when an ultrasound confirms urine in the bladder. The question remains: what is the best method for sterile collection of urine in neonates? In this study, the investigators will try to answer this question by collecting urine from neonates using either ultrasound guided SPA or UC and then comparing the contamination rates between these two methods.

The investigators hypothesize that SPA will result in less contamination of urine samples.

The investigators also hypothesize that there will be more success in obtaining an adequate urine sample (0.5 ml) by SPA, and that there will be no difference in associated complication rates between SPA and UC.

DETAILED DESCRIPTION:
See above and other sections.

ELIGIBILITY:
Inclusion criteria (to be approached for consent):

-All infants who are admitted to the NICU and are not known to have the exclusion criteria listed below at the time of admission

Exclusion criteria (to be approached for consent):

* Antenatal detection or suspicion of genitourinary anomaly including: ambiguous genitalia, hypospadias, posterior urethral valve, anal atresia, exstrophy-epispadias complex, and oligohydramnios secondary to probable genitourinary anomaly(e.g. renal agenesis, multicystic kidney disease)
* Antenatal hydrops
* Antenatally detected abdominal wall defect or abdominal masses
* Antenatally detected grossly dilated bowel loops
* Congenital abdominal skin lesion over the SPA puncture site

Inclusion criteria (prior to randomization):

-All infants who are greater than 72 hours of age, who are being investigated for a possible UTI, and have been consented will be eligible for randomization

Exclusion criteria (prior to randomization):

* Oliguria (<0.5 cc/kg/hr) or anuria over the 8 hours prior to attempted urine collection
* Skin infection over the SPA puncture site
* Distension or enlargement of abdominal viscera (e.g. grossly dilated loops of bowel or massive organomegaly)
* Active Necrotizing enterocolitis (Bell stage II or more)
* Uncorrected thrombocytopenia (platelets < 50 x 10 6) or bleeding diathesis
* Post-abdominal surgery
* Large inguinal hernia
* Current pre-existing indwelling catheter

Ages: 72 Hours to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of contaminated urine samples per SPA and UC | up to 2 years
  For SPA samples, urine contamination will be defined as the growth of two or more micro-organisms (any number of colonies per each microorganism) or the growth of Candida species plus growth of any other microorganism.
  For UC samples, urine contamination will be defined as the growth of two or more micro-organisms (any number of colonies per each microorganism) or any growth <10^4 colony forming unit(CFU)/ml or the growth of Candida species plus growth of any other microorganism.
  The different cut-off used for contamination between UC and SPA samples stems from the fact that the UC procedure is not sterile in the neonatal population.
  Note that a bacterial load of <10^3 CFU/mL (e.g. 10^1 or 10^2 CFU/mL) does not grow in the media of either laboratory where our study samples are being cultured.
  Further sensitivity analyses will be performed on this outcome measure.

SECONDARY OUTCOMES:
Success rates of obtaining urine by SPA versus UC | up to 2 years
  Successful withdrawal of urine is defined as obtaining 0.5ml of urine during an attempt at SPA or UC. This is the quantity required by our laboratory for urine culture.
Time to perform the respective procedures | up to 2 years
  Start time will be recorded as initiation of sterile preparation of the skin. Finish time will be recorded as removal of SPA needle or UC catheter. In the event that the catheter is to remain indwelling, finish time will be recorded as the cessation of sample collection for culture
Complication rates of SPA versus UC | up to 2 years
  UC complications
  * macroscopic hematuria within 48 hours after the procedure including the first void.
  * urinary retention (completely dry diaper with the presence of a distended bladder based on palpation and/or percussion) within the first 4 hours after the procedure.
  SPA complications
  * macroscopic hematuria within 48 hours after the procedure including the first void after the procedure.
  * bowel perforation defined as the aspiration of stool contents or clinical and radiographic signs present within 4-6 hrs after the procedure.
  * suprapubic hematoma or abscess occurring within 1 week after the procedure
  * clinical peritonitis based on the new presence of some or all of the following: fever, tachycardia, absent bowel sounds, abdominal distension, guarding, rigidity or tenderness, and vomiting occuring within 72 hours after the procedure.
Contamination rates of SPA versus UC (excluding clean catch urine) | up to 2 years
  Since the investigators will collect a clean catch urine sample if the randomly assigned infant passes urine spontaneously during a UC attempt but not during SPA attempt, the investigators will compare the contamination rates per UC versus SPA with the exclusion of clean catch samples to ensure pure comparison between the two procedures.
Number of attempts per procedure | up to 2 years
  For UC: each time a urinary catheter is introduced through the foreskin or the urethral meatus, this will be considered one attempt.
  For SPA: each time the skin is punctured by the needle, this will be considered one attempt. This allows for an attempt to include redirection of the needle as long as it remains beneath the skin.
  We will be assessing for a procedural learning curve through this outcome measure and the data recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P Moore, MD, Principal Investigator — Children's Hospital of Eastern Ontario; Ottawa Hospital; University of Ottawa
Locations (2):
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Ottawa Hospital - General campus, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No